CLINICAL TRIAL: NCT06188000
Title: Efficacy of Extra Virgin Olive Oil (EVOO) Supplementation on Serum COX-2, Malondialdehyde, TNF-alpha, and Hand-Foot Syndrome Incidence in Patients With Capecitabine
Brief Title: Efficacy of Extra Virgin Olive Oil (EVOO) Supplementation on Hand-Foot Syndrome Incidence in Patients With Capecitabine
Acronym: EVOO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Universitas Sriwijaya (Other)
Responsible Party: Principal Investigator, Yenny Andayani, Head of Hematology and Clinical Oncology Division, Department of Internal Medicine, Universitas Sriwijaya/Mohammad Hoesin General Hospital, Universitas Sriwijaya
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 069/kepkrsmh/2022
Record Dates: First submitted 2023-03-14; First posted 2024-01-03 (Actual); Last update posted 2024-01-03 (Actual); Status verified 2024-01

CONDITIONS: Hand and Foot Skin Reaction; Hand and Foot Syndrome; Capecitabine
MeSH Terms: conditions — Hand-Foot Syndrome | interventions — Olive Oil

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Extra Virgin Olive Oil (Experimental): The patients was given a capsule contained extra virgin olive oil 15 milliliters twice a day.
  Interventions: Dietary Supplement: Extra Virgin Olive Oil
- Olive Oil (Active Comparator): The patients was given a capsule contained olive oil 15 milliliters twice a day.
  Interventions: Dietary Supplement: Olive Oil
- Placebo (Placebo Comparator): The patients was given an empty capsule twice a day.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Extra Virgin Olive Oil — The patients was given extra virgin olive oil, an unrefined (not processed with chemicals or heat) for of olive oil
  Other Names: EVOO
  Arms: Extra Virgin Olive Oil
Dietary Supplement: Olive Oil — The patients was given olive oil.
  Arms: Olive Oil
Dietary Supplement: Placebo — The patients was given empty capsule
  Arms: Placebo

SUMMARY:
The study was aimed to evaluate the efficacy of extra virgin olive oil (EVOO) supplementation compared to placebo to prevent HFS by observing changes in serum COX 2, malondialdehyde (MDA), and TNF α levels in breast cancer and colorectal cancer patients undergoing capecitabine chemotherapy. Current study was designed as a single-center prospective randomized clinical trial. The patients were Stage III or Stage IV colorectal and breast cancer patients receiving capecitabine-based chemotherapy who enrolled in the trial voluntarily. All patients were divided randomly into three groups treated with EVOO, olive oil, or placebo. The incidence of hand foot syndrome was documented. The serum COX 2, malondialdehyde (MDA), and TNF α levels before and after chemotherapy was documented.

ELIGIBILITY:
Inclusion Criteria:

* Patients pathologically and clinically diagnosed with III or IV stadium of breast cancer or colorectal cancer.
* fully recovered after curative resection within 8 weeks
* receive adjuvant capecitabine based chemotherapy

Exclusion Criteria:

* did not meet the eligibility criteria for chemotherapy
* had previous allergy with capecitabine or olive oil

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2024-02-01 (Estimated); Study Completion 2024-02-20 (Estimated)

PRIMARY OUTCOMES:
Hand Foot Syndrome | 3 cycle of chemotherapy (63 days)
  Patients was documented for hand and foot syndrome using WHO criteria. There were 4 grade assessed by patient symptoms of tingling or burning or painful sensation, palmar or plantar erythema or desquamation, and/or ulceration.
Serum COX-2 Concentration | 3 cycle of chemotherapy (63 days)
  Serum COX-2 Concentration
Serum malondialdehyde concentration | 3 cycle of chemotherapy (63 days)
  Serum malondialdehyde ceoncentration
Serum Tumor Necrosis Factor Alpha Concentration | 3 cycle of chemotherapy (63 days)
  Serum Tumor Necrosis Factor Alpha Concentration

CONTACTS AND LOCATIONS:
Locations (1):
- Rumah Sakit Mohammad Hoesin, Palembang, South Sumatera, Indonesia

IPD SHARING:
Plan to Share IPD: No
The data will be shared after the completion of the study and has been subjected to the consent of the individual patients

REFERENCES:
- [Background] Huang XZ, Chen Y, Chen WJ, Zhang X, Wu CC, Wang ZN, Wu J. Clinical evidence of prevention strategies for capecitabine-induced hand-foot syndrome. Int J Cancer. 2018 Jun 15;142(12):2567-2577. doi: 10.1002/ijc.31269. Epub 2018 Feb 2. PMID 29355976
- [Background] Deng B, Sun W. Herbal medicine for hand-foot syndrome induced by fluoropyrimidines: A systematic review and meta-analysis. Phytother Res. 2018 Jul;32(7):1211-1228. doi: 10.1002/ptr.6068. Epub 2018 Apr 16. PMID 29682836
- [Background] Elyasi S, Rasta S, Taghizadeh-Kermani A, Hosseini S. Topical henna and curcumin (Alpha(R)) ointment efficacy for prevention of capecitabine induced hand-foot syndrome: A randomized, triple-blinded, placebo-controlled clinical. Daru. 2022 Jun;30(1):117-125. doi: 10.1007/s40199-022-00438-8. Epub 2022 Mar 23. PMID 35320555
- [Result] Zhang RX, Wu XJ, Wan DS, Lu ZH, Kong LH, Pan ZZ, Chen G. Celecoxib can prevent capecitabine-related hand-foot syndrome in stage II and III colorectal cancer patients: result of a single-center, prospective randomized phase III trial. Ann Oncol. 2012 May;23(5):1348-1353. doi: 10.1093/annonc/mdr400. Epub 2011 Sep 22. PMID 21940785
- [Result] Yap YS, Kwok LL, Syn N, Chay WY, Chia JWK, Tham CK, Wong NS, Lo SK, Dent RA, Tan S, Mok ZY, Koh KX, Toh HC, Koo WH, Loh M, Ng RCH, Choo SP, Soong RCT. Predictors of Hand-Foot Syndrome and Pyridoxine for Prevention of Capecitabine-Induced Hand-Foot Syndrome: A Randomized Clinical Trial. JAMA Oncol. 2017 Nov 1;3(11):1538-1545. doi: 10.1001/jamaoncol.2017.1269. PMID 28715540